CLINICAL TRIAL: NCT03236051
Title: Multimodal Analgesia in Laparoscopic Radical Gastrectomy With Gastric Cancer: a Multi-center Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: JIANG Zhi-Wei (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, JIANG Zhi-Wei, Vice director of Research Institute of General Surgery, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016HR1116
Record Dates: First submitted 2017-07-26; First posted 2017-08-01 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; gastrectomy; multimodal analgesia; parecoxib
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a randomized, parallel, controlled, open study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multimodal analgesia (Experimental): Patients received multimodal analgesia after laparoscopic gastrectomy .
  Interventions: Procedure: Multimodal analgesia
- PCIA analgesia (Active Comparator): Patients received PCIA analgesia after laparoscopic gastrectomy.
  Interventions: Procedure: PCIA analgesia

INTERVENTIONS:
Procedure: Multimodal analgesia — Multimodal analgesia is the name of a procedure or program. Multimodal analgesia doesn't mean different interventions are used. Patients in this group need receive this analgesia program (procedure) instead of one analgesic drug or technology. The program consists of incision infiltration with ropivacaine, intravenous injection of parecoxib, and oral administration of oxycodone/paracetamol mixture.
  Arms: multimodal analgesia
Procedure: PCIA analgesia — PCIA analgesia:patient-controlled intravenous analgesia with tramadol.
  Arms: PCIA analgesia

SUMMARY:
The study is aimed to explore the effects of multimodal analgesia consisting of ropivacaine's wound infiltration, parecoxib's intravenous injection and oxycodone-acetaminophen tablets' oral administration on postoperative pain and rehabilitation after laparoscopic radical gastrectomy for patients with gastric cancer.

DETAILED DESCRIPTION:
Postoperative pain attracts the attention of surgeons, and optimal postoperative pain management contributes to reducing complications and accelerating postoperative rehabilitation. Traditionally, the opioids were used for postoperative pain control. However, the opioids may increase the time to recover bowel function and lead to postoperative ileus. Multimodal analgesia is recommended in recent years, but studies on multimodal analgesia after gastrectomy are scarce. In this study, we introduced a multimodal analgesia strategy consisting of incision infiltration with ropivacaine, intravenous injection of parecoxib, and oral administration of an oxycodone/paracetamol mixture and evaluated the effects of this strategy compared with PCIA analgesia which is used widely for pain after gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Requirements of informed consent and assent of participant, parent or legal guardian as applicable.
2. Patients underwent laparoscopic radical gastrectomy under general anesthesia and between the age of 18 and 75 years old without considering sex.
3. American Society of Anesthesiologists (ASA) physical status I-III.
4. Participants can follow the drug doses and visit plan

Exclusion Criteria:

1. Patients certified by a doctor that doesn't fit to participate in this study.
2. Patients allergic to opioids, sulfas, parecoxib, non-steroidal drugs, acetaminophen, tramadol etc..
3. Patients with ischemic heart disease, cerebrovascular disease and peripheral vascular disease, or their cardiac function > II (NYHA) patients, patients received coronary artery bypass grafting (CABG) recently, and patients with severe hypertension (systolic pressure≥180mmHg or diastolic pressure≥110mmHg).
4. Patients with gastric cancer with distant metastasis.
5. Patients with severe infection, respiratory dysfunction, coagulation disorders, severe liver and renal dysfunction (Child - Pugh≥ 10; creatinine clearance < 25 ml/min).
6. Patients with suspect or have a history of drug abuse.
7. Pregnancy and lactation women, or have a pregnancy plan within a month after the test of the subjects (also including male participants).
8. Sponsors or researchers directly involved in the testing or their family members.
9. Patients with conversion, palliative resection.
10. Patients with chronic pain（NRS≥3）or using opioids or NSAIDs before surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2017-02-10 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-08-30 (Estimated)

PRIMARY OUTCOMES:
Numeric rating scales (NRS) score with 24 hours after the surgery | 1 day
  pain evaluation

SECONDARY OUTCOMES:
NRS score after 24 hours postoperatively | 1 week
  pain evaluation
Number of remedial treatment | 1 week
  pain evaluation
Time to first flatus | 1 week
  Bowel function recovery
Time to first off-bed activity | 1 week
  Postoperative activity
Time of off-bed activity per day | 1 week
  Postoperative activity
Length of off-bed activity per day | 1 week
  Postoperative activity
Time to first semi-liquid diet | 1 week
  Bowel function recovery
Postoperative length of stay | 1 month
  postoperative length of stay
C-reactive protein (CRP) | 1 week
  Inflammatory indicators
interleukin-6 (IL-6) | 1 week
  Inflammatory indicators
Albumin | 1 year
  Nutritional status
Total protein | 1 year
  Nutritional status
Prealbumin | 1 year
  Nutritional status

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Wei JIANG, Ph.D., Principal Investigator — Jinling Hospital, Medical School of Nanjing University; Jian ZHAO, Ph.D., Study Director — Jinling Hospital, Medical School of Nanjing University; Gang WANG, Ph.D., Study Director — Jinling Hospital, Medical School of Nanjing University; Jiang LIU, M.D., Study Director — Jinling Hospital, Medical School of Nanjing University
Locations (2):
- China (2):
  - Jinling Hospital, Medical School of Nanjing University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No